CLINICAL TRIAL: NCT05056467
Title: Labor Induction Versus Expectant Management in High-risk Women for Preeclampsia
Brief Title: Labor Induction in Preeclampsia High-risk Women
Acronym: FORECAST-IOL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Hanoi Obstetrics and Gynecology Hospital (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Angel Women and Children Hospital (Unknown); Rumah Sakit Anak dan Bunda Harapan Kita (Unknown); National University Hospital, Singapore (Other); Taiji Clinic, Taiwan (Unknown); Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Chiu Yee Liona Poon, Professor (Clinical), Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021.249
Record Dates: First submitted 2021-09-20; First posted 2021-09-24 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Pre-Eclampsia; Induction of Labor
Keywords: aspirin; biomarker; blood pressure; hypertension; mean arterial pressure; placental growth factor; pre-eclampsia; prediction; uterine artery pulsatility index; induction of labor
MeSH Terms: conditions — Pre-Eclampsia; Hypertension | interventions — Labor, Induced

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IOL (Experimental): Preeclampsia High-risk Women schedule labor induction at 39 weeks of gestation
  Interventions: Procedure: Induction of Labor
- Expectant Management (No Intervention): Preeclampsia High-risk Women under expectant management

INTERVENTIONS:
Procedure: Induction of Labor — Induction of Labor at 39 weeks of gestation
  Arms: IOL

SUMMARY:
Preeclampsia (PE) is one of the leading causes of maternal and perinatal morbidity and mortality. This pregnancy-specific disorder poses to both pregnant women and their offspring an increased risk of immediate and long-term health problems. The study team is conducting a study entitled "FORECAST" (Implementation of First-trimester Screening and preventiOn of pREeClAmpSia Trial) and established the infrastructure for the first-trimester "screen and prevent" program for preterm PE. However, there is no established evidence regarding the benefit of scheduled labor induction versus expectant management among women identified as high-risk for PE with uncomplicated pregnancy at term. The investigators postulate that induction of labor at 39 weeks' gestation may possibly be an effective intervention to reduce placental complications in women with uncomplicated pregnancy by 39 weeks at high-risk PE women.

ELIGIBILITY:
Inclusion Criteria:

* Age no less than 18 years
* Singleton pregnancy with cephalic presentation and no contraindication to vaginal delivery
* Live fetus
* Screened high-risk for PE
* Informed and written consent

Exclusion Criteria:

* Multiple pregnancy
* Pregnant women who plan to have Cesarean delivery
* Pregnancies complicated by the major fetal abnormality
* Women who are severely ill, those with learning difficulties, or serious mental illness
* Pregnant women with medical, obstetric, or fetal complications or any other indications for delivery before 39 weeks' gestation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 825 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
the rate of adverse placental outcomes | At Delivery
  To compare the difference in the rate of adverse placental outcomes (PE, gestational hypertension (GH), SGA, stillbirth, perinatal death, placental abruption) in the induction of labor group with the expectant management group.

SECONDARY OUTCOMES:
the rate of adverse maternal outcomes | 6 weeks Postpartum
  To compare the difference in the rate of maternal secondary outcomes including composite outcomes of the following: Cesarean delivery/indication for Cesarean delivery, operative vaginal delivery, indication for operative vaginal delivery, uterine incisional extensions during Cesarean delivery, chorioamnionitis, third-degree or fourth-degree perineal laceration, postpartum hemorrhage, postpartum infection, venous thromboembolism, number of hours in the labor and delivery unit, length of postpartum hospital stay, admission to the intensive care unit, and maternal death, between the induction of labor group and the expectant management group.
the rate of adverse neonatal outcomes | 28 days after birth
  To compare the difference in the rate of neonatal secondary outcomes including the composite outcomes of the following: perinatal death or severe neonatal complications and consisted of one or more of the following during the antepartum or intrapartum period or during the delivery hospitalization between the induction of labor group and the expectant management group.

CONTACTS AND LOCATIONS:
Locations (8):
- China (2):
  - Angel Women's and Children's Hospital, Chengdu
  - The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing
- Prince of Wales Hospital, Hong Kong, Hong Kong
- Harapan Kita Hospital, Jakarta, Indonesia
- National University Hospital, Singapore, Singapore
- Taiji Clinic, Taipei, Taiwan
- Siriraj Hospital, Bangkok, Thailand
- Hanoi Obstetrics & Gynecology Hospital, Hanoi, Vietnam